CLINICAL TRIAL: NCT00834067
Title: A Relative Bioavailability Study of Moexipril HCl/Hydrochlorothiazide 15/25 mg Tablets Under Non-Fasting Conditions
Brief Title: Moexipril HCl/Hydrochlorothiazide 15/25 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B036544
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Moexipril HCl/hydrochlorothiazide 15/25 mg tablets
- 2 (Active Comparator)
  Interventions: Drug: UNIRETIC® 15/25 mg tablets

INTERVENTIONS:
Drug: Moexipril HCl/hydrochlorothiazide 15/25 mg tablets — 1 x 15/25 mg
  Arms: 1
Drug: UNIRETIC® 15/25 mg tablets — 1 x 15/25 mg
  Arms: 2

SUMMARY:
The objective of this study is to compare the relative bioavailability of moexipril HCl/ hydrochlorothiazide 15/25 mg tablets (manufactured and distributed by TEVA Pharmaceuticals USA) with that of UNIRETIC® 15/25 mg tablets (Schwartz Pharma) in healthy, adult, non-smoking subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be non-smokers at least 18 years of age.
* Subjects will have a BMI index (body mass index) of 30 or less.

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result not to be significant.
* Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study.
* All subjects will have urine samples assayed for the presence of abuse as part of the clinical laboratory screening procedures and ath check-in each study period. Subjects found to have urine concentrations of any of the tested drug will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken an investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives anytime during the 180 days prior to study dosing or oral hormonal contraceptives with in 14 days of dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.
* Subjects who do not tolerate venipuncture will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Plisco, M.D., Principal Investigator — Gateway Medical Research
Locations (2):
- United States (2):
  - Gateway Medical Research, Inc., Saint Charles, Missouri
  - Bioassay Laboratory, Inc., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Moexipril HCl/HCTZ) First: 15/25 mg Moexipril HCl/Hydrochlorothiazide Tablets test product dosed in first period followed by 15/25 mg Uniretic® Tablets reference product dosed in the second period.
- Reference (Uniretic®) First: 15/25 mg Uniretic® Tablets reference product dosed in first period followed by 15/25 mg Moexipril HCl/Hydrochlorothiazide Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Moexipril HCl/HCTZ) First | Reference (Uniretic®) First
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Washout of 21 Days
Arm/Group | Test (Moexipril HCl/HCTZ) First | Reference (Uniretic®) First
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Second Intervention
Arm/Group | Test (Moexipril HCl/HCTZ) First | Reference (Uniretic®) First
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Moexipril HCl/HCTZ) First | Reference (Uniretic®) First | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 17 | 16 | 33
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  Black | 7 | 2 | 9
  White | 22 | 25 | 47
  Hispanic | 1 | 1 | 2
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma) of Moexipril.
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Moexipril HCl/HCTZ): 15/25 mg Moexipril HCl/Hydrochlorothiazide Tablets test product dosed in either period.
- Reference (Uniretic®): 15/25 mg Uniretic® Tablets reference product dosed in either period.
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng/mL | 14.487 (6.706) | 14.885 (6.018)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 96.7, 90% CI [90.1 to 104] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration) of Moexipril.
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng*h/mL | 35.412 (41.756) | 34.917 (47.077)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 104, 90% CI [99.9 to 108] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity) of Moexipril.
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng*h/mL | 36.651 (43.262) | 35.74 (47.957)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 103, 90% CI [99.7 to 107] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma) of Hydrochlorothiazide.
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng/mL | 150.225 (42.664) | 148.39 (39.83)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101, 90% CI [96 to 106] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration) of Hydrochlorothiazide.
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng*h/mL | 1105.63 (260.669) | 1100.5 (271.834)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101, 90% CI [99.1 to 102] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity) of Hydrochlorothiazide.
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng*h/mL | 1115.905 (259.765) | 1108.329 (271.82)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101, 90% CI [99.4 to 103] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma) of Moexiprilat.
Description: Informational comparison of Cmax values for the metabolite Moexiprilat.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng/mL | 5.512 (3.241) | 5.13 (2.788)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 107, 90% CI [99.8 to 114] — This analysis was for informational purposes only and was not used to establish bioequivalence

8. Secondary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration) of Moexiprilat.
Description: Informational comparison of AUC0-t values for the metabolite Moexiprilat.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng*h/mL | 215.654 (61.545) | 214.286 (69.726)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102, 90% CI [99 to 106] — This analysis was for informational purposes only and was not used to establish bioequivalence

9. Secondary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity) of Moexiprilat.
Description: Informational comparison of AUC0-inf values for the metabolite Moexiprilat.
Time Frame: Blood samples collected over a 192 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Moexipril HCl/HCTZ) | Reference (Uniretic®)
Number analyzed (Participants) | 59 | 59
ng*h/mL | 376.814 (144.282) | 379.994 (184.852)
Statistical Analysis 1: Comparison: Test (Moexipril HCl/HCTZ) vs Reference (Uniretic®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 103, 90% CI [98.1 to 108] — This analysis was for informational purposes only and was not used to establish bioequivalence

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.